CLINICAL TRIAL: NCT05866107
Title: Effectiveness and Feasibility of Self-Monitoring for Weight Management in Individuals With Mental Disorders Using Digital Intervention ("SWIM" Trial)
Brief Title: App and Body Fat Scale in the Management of Overweight Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Le Xiao, Chief Physician, Beijing Anding Hospital, Capital Medical University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MISP#100150
Record Dates: First submitted 2023-03-06; First posted 2023-05-19 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia; Bipolar Disorder; Metabolic Syndrome; Overweight and Obesity
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Metabolic Syndrome; Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Batch 1 (Intervention from Month 3) (Experimental): 3 clinical units (clusters) receiving the combined digital and multidisciplinary intervention starting at Month 3. Each unit includes approximately 34 patients (total n=102) with schizophrenia or bipolar disorder.
  Interventions: Device: Effectiveness and Feasibility of Self-Monitoring for Weight Management in Individuals with Mental Disorders Using Digital Intervention ("SWIM" trial)
- Batch 2 (Intervention from Month 5) (Experimental): 3 clinical units (clusters) receiving the same intervention starting at Month 5. Each unit includes approximately 34 patients (total n=102) with schizophrenia or bipolar disorder.
  Interventions: Device: Effectiveness and Feasibility of Self-Monitoring for Weight Management in Individuals with Mental Disorders Using Digital Intervention ("SWIM" trial)

INTERVENTIONS:
Device: Effectiveness and Feasibility of Self-Monitoring for Weight Management in Individuals with Mental Disorders Using Digital Intervention ("SWIM" trial) — Participants receive a digital-behavioral intervention via Huawei Health App and smart scale:
  1. Weekly weigh-ins (auto-synced)
  2. Dietary logging (≥3x/week) with calorie-deficit targets
  3. Biweekly exercise plans (150-300 min/week)
  4. Weekly motivational messages
  Implementation:
  Staggered rollout: Batch 1 (Month 3-6), Batch 2 (Month 5-6). Includes 2-week training. Effectiveness monitored via app metrics and adherence. Routine care maintained.

SUMMARY:
This study tests whether using a health app (Huawei Health) and a smart body fat scale can help overweight patients with schizophrenia or bipolar disorder lose weight and stay engaged in their health.

What We're Testing:

1. Patients who use the app and scale for 4 months (Group 1) will lose more weight than those who use them for 2 months (Group 2).
2. Patients who track their weight, diet, and exercise regularly (≥3 times/week) will lose more weight than those who don't.
3. Seeing weight loss results may motivate patients to keep using the app and scale.

How It Works:

Patients weigh themselves weekly with the scale (auto-syncs to the app) and upload dietary log in Huawei Health app. The app will gives personalized diet/exercise tips and tracks progress. Doctors and nutritionists provide extra support through messages.

Goal:

To see if this digital tool + professional support combo works better for long-term weight management.

DETAILED DESCRIPTION:
The investigators will recruit the patients diagnosed with schizophrenia or bipolar disorder from Beijing Anding Hospital. Participants will use a mobile phone app (Huawei Health) to collect data on daily activities and calorie consumption. The smart body fat scale with high-precision weighing chip (Huawei Scale 2pro) will be used to collect heart rate, weight, BMI, body type, basal metabolic rate, fat rate, fat free body weight, skeletal muscle mass, bone salt content, visceral fat grade, body water (%), body protein rate and body composition, and all data will be uploaded to the app. Participants could also record their daily dietary intake (for calculation of calorie intake) in the health app. This is a 6-month, single-center, stepped wedge-shaped cluster randomized study. It is planned to recruit 204 overweight subjects from 6 units from Beijing Anding Hospital. The six clinical units comprise four inpatient wards, one day rehabilitation unit, and one outpatient department. All units (clusters) were randomly allocated to two batches (3 units each) using a computer-generated sequence. Batch 1 received the intervention from Month 3 to Month 6, while Batch 2 started from Month 5 to Month 6 (total study duration: 6 months). All units underwent baseline observation during Months 1-2, followed by a 2-week transition period for training. All clusters follow usual care prior to their assigned intervention period, with months 1-2 serving as baseline control and months 7-8 for full-intervention observation across all units. Each unit operates as an independent intervention cluster with dedicated staff teams and unit-specific WeChat-based communication groups. Intervention materials, reinforcement messages, counseling content, and technical support are synchronized with each cluster's assigned timeline. Clinical staff will be trained on intervention delivery, digital tool usage, and adherence protocols and are required to adhere strictly to the scheduled rollout sequence. Monitoring and supervision mechanisms will be implemented to track adherence, engagement, and protocol compliance in real-time. Each cluster undergoes a two-week pre-implementation transition period for device distribution, app installation, and training. The intervention combines self-weighing using using smart body fat scale, dietary logging, exercise management, and behavioral reinforcement. Behavioral reinforcement includes weekly personalized feedback messages and real-time alerts for missed self-monitoring via WeChat messages. We assess clinical, functional, and subjective outcomes at baseline and monthly intervals. Socio-demographic and clinical characteristics (age, sex, education, income, medical history) are extracted from EHRs. Body composition metrics (BMI, body fat percentage, etc.) are automatically recorded during weigh-ins. Subjective outcomes will be collected using validated scales at Month 1,2,3 and 6. Smart scale pairing success rate and weekly weigh-in adherence will be used to assess protocol feasibility. To capture user perspectives on mobile app and weighing smart scale, we will conduct 30-minute semi-structured interviews with 30 purposely selected participants (stratified by adherence and diagnosis), exploring app usability, behavioral impacts, and improvement suggestions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old, no gender restriction.
* According to ICD-10 to diagnose bipolar disorder or schizophrenia, the researcher judges that the patient is currently in remission, or the condition is stable and can cooperate with the research.
* Currently using at least one antipsychotic or mood stabilizer (e.g. lithium, magnesium valproate, sodium valproate, lamotrigine).
* Currently overweight or obese (body mass index ≥ 24kg/m2) and willing to use health app and smart scales to lose weight.
* The education level of primary school or above, able to understand the content of the scale, and be able to use smart phone proficiently.
* Understand and voluntarily participate in this study, and sign the informed consent form.

Exclusion Criteria:

* Plan to lose weight by other methods during the study period (such as dieting, inducing vomiting, taking diet pills, surgery).
* Self-reported weight loss ≥ 7% in the past 6 months.
* Weight over 150 kg.
* Other secondary obesity (such as hypothyroidism, Cushing's syndrome, hypothalamic obesity, etc.).
* Currently pregnant, lactating, < 6 months postpartum or planning to become pregnant during the study period.
* Self-reported cardiac discomfort or chest pain during activity or at rest.
* There is a serious medical condition, and the researchers believe that there may be safety risks when participating in sports.
* Be unable to walk 30 minutes without stopping.
* There are problems that may affect compliance with the protocol (eg, end-stage disease, planning to move travel to the field, history of substance abuse, other uncontrolled or untreated medical conditions);
* Any other conditions deemed inappropriate by the investigator.

Participants include approximately 50% with schizophrenia and 50% with bipolar disorder, distributed across all clusters.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percent weight loss | At the end of Months 1, 2, 3, and 6
  Proportion of body weight lost, assessed via smart scale synced with app. Factors distinguish those who do/don't lose weight is detected by using machine learning.
Adherence to self-monitoring | At the end of Months 1, 2, 3, and 6
  Number of days per week participants complete self-weighing, dietary logging and follow up visits.

SECONDARY OUTCOMES:
Longitudinal adherence to self-monitoringcompliance to app + scale protocol and the participants who have bad compliance is compared by percent weight loss. | At the end of Months 1, 2, 3, and 6
  Adherence measured as self-monitoring days per week, assessed monthly across the 6-month study.
Weight loss by adherence level | At the end of Months 1, 2, 3, and 6
  Comparison of percent weight loss between high- and low-adherence groups.
Association between adherence and weight loss | At the end of Months 1, 2, 3, and 6
  Independent variables include diagnosis, treatment, baseline weight, self-monitoring adherence, %WL from the previous month (e.g., %WL at the end of month 2 predicted self-monitoring during month 3), and the interaction between condition and %WL.
Prediction of future adherence by prior weight loss | At the end of Months 1, 2, 3, and 6
  Generalized linear mixed models will test whether weight loss in a given month predicts adherence in the following month.

CONTACTS AND LOCATIONS:
Overall Officials: Le Xiao, Study Chair — Capital Medical University
Locations (1):
- Beijing Anding Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data (including demographics, clinical outcomes, and body composition metrics) will be released to participants and referring clinicians upon request
Supporting Information: Study Protocol
Time Frame: Data will be available from 6 months after primary publication for 5 years
Access Criteria: Researchers must submit a proposal to the corresponding author, subject to approval by the ethics committee

REFERENCES:
- [Result] Tek C, Kucukgoncu S, Guloksuz S, Woods SW, Srihari VH, Annamalai A. Antipsychotic-induced weight gain in first-episode psychosis patients: a meta-analysis of differential effects of antipsychotic medications. Early Interv Psychiatry. 2016 Jun;10(3):193-202. doi: 10.1111/eip.12251. Epub 2015 May 12. PMID 25962699
- [Result] Dayabandara M, Hanwella R, Ratnatunga S, Seneviratne S, Suraweera C, de Silva VA. Antipsychotic-associated weight gain: management strategies and impact on treatment adherence. Neuropsychiatr Dis Treat. 2017 Aug 22;13:2231-2241. doi: 10.2147/NDT.S113099. eCollection 2017. PMID 28883731
- [Result] Brockmann AN, Eastman A, Ross KM. Frequency and Consistency of Self-Weighing to Promote Weight-Loss Maintenance. Obesity (Silver Spring). 2020 Jul;28(7):1215-1218. doi: 10.1002/oby.22828. Epub 2020 May 21. PMID 32437055
- [Result] Patel ML, Wakayama LN, Bennett GG. Self-Monitoring via Digital Health in Weight Loss Interventions: A Systematic Review Among Adults with Overweight or Obesity. Obesity (Silver Spring). 2021 Mar;29(3):478-499. doi: 10.1002/oby.23088. PMID 33624440
- [Result] Cheatham SW, Stull KR, Fantigrassi M, Motel I. The efficacy of wearable activity tracking technology as part of a weight loss program: a systematic review. J Sports Med Phys Fitness. 2018 Apr;58(4):534-548. doi: 10.23736/S0022-4707.17.07437-0. Epub 2017 May 9. PMID 28488834
- [Result] Suen L, Wang W, Cheng KKY, Chua MCH, Yeung JWF, Koh WK, Yeung SKW, Ho JYS. Self-Administered Auricular Acupressure Integrated With a Smartphone App for Weight Reduction: Randomized Feasibility Trial. JMIR Mhealth Uhealth. 2019 May 29;7(5):e14386. doi: 10.2196/14386. PMID 31144666
- [Result] Flores Mateo G, Granado-Font E, Ferre-Grau C, Montana-Carreras X. Mobile Phone Apps to Promote Weight Loss and Increase Physical Activity: A Systematic Review and Meta-Analysis. J Med Internet Res. 2015 Nov 10;17(11):e253. doi: 10.2196/jmir.4836. PMID 26554314
- [Result] Goldstein SP, Goldstein CM, Bond DS, Raynor HA, Wing RR, Thomas JG. Associations between self-monitoring and weight change in behavioral weight loss interventions. Health Psychol. 2019 Dec;38(12):1128-1136. doi: 10.1037/hea0000800. Epub 2019 Sep 26. PMID 31556659
- [Result] Patel ML, Hopkins CM, Brooks TL, Bennett GG. Comparing Self-Monitoring Strategies for Weight Loss in a Smartphone App: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Feb 28;7(2):e12209. doi: 10.2196/12209. PMID 30816851